CLINICAL TRIAL: NCT01027806
Title: A Randomized Double Blind Controlled Trial on the Effect of Montelukast Treatment in Children With Obstructive Sleep Apnea Syndrome
Brief Title: Effect of Montelukast Therapy in Obstructive Sleep Apnea(OSA) Children
Acronym: 32543
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-008A
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Children; Sleep; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator)
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator)
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — 1 pill per day for 4 months

SUMMARY:
The investigators leading hypotheses are:

* Oral therapy with montelukast may lead to improved sleep study findings in children with mild to moderate Obstructive Sleep Apnea Syndrome (OSAS) who require surgical removal of adenoids and tonsils for OSAS.
* A significant proportion of the children with OSAS treated with montelukast will show reduced severity of OSAS, and this will remove the need for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for inclusion in the study will be symptomatic snoring children >2 years of age and < 10 years of age, who snore and have an apnea hypopnea index (AHI) >2/hrTST (hour total sleep time), and in whom T&A is therefore contemplated. Also among these, we will include children referred for evaluation for snoring who have a history of allergic rhinitis.

Exclusion Criteria:

* Exclusion criteria will include: Hypersensitivity to montelukast, immunodeficiency or immunosuppressant therapy, craniofacial, neuromuscular, syndromic or defined genetic abnormalities, acute upper respiratory tract infection, systemic corticosteroid therapy or antibiotic therapy in the 2 weeks previous to the study, and children who already had adenotonsillectomy. In addition, children chronically receiving oral antihistamine preparations or nasal decongestants will be required to continue using these medications throughout the duration of the study. Patients receiving immunotherapy will continue on the same regimen without escalation of dose and frequency throughout the duration of the study. In addition, patients with severe OSA who in the opinion of their treating physicians require early surgical intervention for their OSA will be excluded from eligibility to the study.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leila Gozal, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast: Montelukast: 1 pill per day for 16 weeks
- Placebo: Placebo: 1 pill per day for 16 weeks
Period: Overall Study
Arm/Group | Montelukast | Placebo
Started | 32 | 32
Completed | 28 | 29
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: Patients who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (2.5) | 5.6 (2.4) | 5.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 12 | 24
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Children Experiencing a Reduction in Apnea-Hypopnea Index (API) From Baseline (Before Treatment) to After Treatment.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 28 | 29
Participants
  Reduction in AHI | 20 | 2
  No reduction in AHI | 8 | 27
Statistical Analysis 1: Comparison: Montelukast vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 2/28 | 3/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Montelukast (N=28) | Placebo (N=29)
Headache (General disorders) | 1 | 1
Nausea (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No